CLINICAL TRIAL: NCT00728351
Title: A Multicenter, Double-blind, Randomized Study to Compare the Efficacy of 24 Weeks Treatment With Fixed Combination Therapy of Vildagliptin and Metformin (25/1000 mg Bid) Versus Metformin Monotherapy (1000 mg Bid) in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy.
Brief Title: Efficacy and Safety of Fixed Combination Therapy of Vildagliptin and Metformin (25/1000 mg Bid) in Patients With Type 2 Diabetes Inadequately Controlled With Prior Metformin Monotherapy (HbA1c 7.0-9.5%)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLMF237A2309
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes, vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin + metformin (Experimental)
  Interventions: Drug: vildagliptin + metformin
- metformin (Active Comparator)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: vildagliptin + metformin
  Arms: vildagliptin + metformin
Drug: metformin — 1000 bid metformin
  Arms: metformin

SUMMARY:
The present study is designed to evaluate the efficacy and safety of fixed combination therapy of vildagliptin and metformin (25/1000 mg bid) in patients with type 2 diabetes inadequately controlled with prior metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of T2DM treated with Metformin

Exclusion Criteria:

* FPG >= 260 mg/dL (14.4mmol/L)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction after 24 weeks of treatment in patients with T2DM inadequately controlled with metformin monotherapy | 24 weeks

SECONDARY OUTCOMES:
FPG reduction | 24 weeks
Safety and tolerability | 24 weeks
Body weight change from baseline | 24 weeks
Changes in the fasting lipid profile | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (61):
- United States (14):
  - Pine Bluff, Arkansas
  - Long Beach, California
  - Denver, Colorado
  - Bangor, Maine
  - Billings, Montana
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Trenton, New Jersey
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Uniontown, Pennsylvania
  - Taylors, South Carolina
  - Houston, Texas
  - Norfolk, Virginia
  - Wenatchee, Washington
- France (3):
  - Cabinet d'Endocrinologie-Maladies Métaboliques, Annecy
  - Service Endocrinologic & Metabolisme, Paris
  - Polycliniques des minguettes, Vénissieux
- Germany (16):
  - Hausärztliche Praxis, Aschaffenburg
  - Klinische Forschung Berlin Mitte GmbH, Berlin
  - AVK, Berlin
  - Gemeinschaftspraxis, Celle
  - Malteser KM, Duisburg
  - Untertrintroper Hausarztzentrum, Essen
  - Gefrees
  - Diabeteszentrum Billstedt/Horn, Hamburg
  - Diabetologische Schwerpunktpraxis, Hamburg
  - St. Elisabeth Krankenhaus Leipzig, Leipzig
  - Diabetes-Schwerpunktpraxis Studienambulanz, Leipzig
  - Institut für Diabetes-forschung Münster, Münster
  - Praxis Dr. Alawi, Saarlouis
  - DDT, Siegen
  - Diabetologische Schwerpunktpraxis, Sinsheim
  - Praxis, Wangen
- Hungary (12):
  - Europ-Med Orvosi Szolgaltato Kft, Budaörs
  - Synexus Magyarorszag, Budapest
  - Uzsoki Hospital, Budapest
  - Budapest
  - Kenezy Hospital, Debrecen
  - Gyngyosi Korhaz Kft, Gyöngyös
  - Petz Aladar County, Győr
  - Selye Janos Korhaz es Rendelointezet, Komárom
  - DIAPED Kft., MRC, Meggyesalja U.
  - Josa Andras Teaching Hospital, Nyíregyháza
  - Vas Megyei Markuscvszky Lajos Korhaz, Szombathely
  - Zala County Hospital, Zalaegerszeg
- Poland (16):
  - NZOZ Specjalistyczny Ośrodek Internistyczno - Diabetologiczny Białystok, Bialystok
  - Gdanska Poradnia Cukrzycowa, Gdansk
  - Gabinet Kardiologiczny Mediplus, Gdynia
  - NZOZ "Esculap" S.C., Gniewkowo
  - SZPZOZ Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki
  - NZOZ Terapia Optima, Katowice
  - Instytut Cantrum Zdrowia Matki Polki, Lodz
  - NZOZ Special-Med, Lublin
  - Szspital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Ponza, Poznan
  - Lecznica Prosen-SMO NZOZ, Warsaw
  - Centrum Leczenia Chorob Cywilizacyjnych, Warsaw
  - NZCZ Regionalna Poradnia Diabetologiczna, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny NR 1 im. Prof. Stanislawa Szysko SAM, Zabrze
  - Poradnia Diabetologiczna, Zespol Opieki Zdrowotnej w Leczycy, Łęczyca
  - Zespół Opieki Zdrowotnej w Łęczycy, Poradnia Diabetologiczna Łeczyca, Łęczyca

REFERENCES:
- See also: Click here for more information on the clinical study — http://www.novartisclinicaltrials.com
- See also: Results for CLMF237A2309 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3860